CLINICAL TRIAL: NCT06856057
Title: Improving Quality of Life and Behavioral Health Service Access for Caregivers and Young Children After Pediatric Traumatic Injury
Brief Title: Improving Behavioral Health for Caregivers and Children After Pediatric Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Leigh Ridings, Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00138482; 1R01HD117024-01 (NIH)
Record Dates: First submitted 2025-02-11; First posted 2025-03-04 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Quality of Life; PTSD; Depression Not Otherwise Specified; Child Externalizing Behavior
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced usual care (EUC) (No Intervention): Educational packet includes behavioral health education for children and families after pediatric traumatic injury(PTI).
- Caregivers' Aid to Accelerate Recovery after pediatric Emergencies (CAARE) (Experimental): CAARE provides bedside screening and education, digital health tools to help caregivers track and manage emotional and behavioral recovery, and timely follow-up to facilitate screening and referrals (if needed). The 4 steps are: (1) a brief bedside intervention for caregivers and children with positive acute stress risk screens designed to provide coping skills and reduce distress; (2) technology resources including (a) a text message-based tool to facilitate symptom self-monitoring and (b) an mHealth application with embedded learning, coping skills, and service locator tools; (3) a 30-day behavioral health screening, and (4) referral to evidence-based treatment for children and caregivers with positive screens.
  Interventions: Behavioral: Caregivers' Aid to Accelerate Recovery after pediatric Emergencies (CAARE)

INTERVENTIONS:
Behavioral: Caregivers' Aid to Accelerate Recovery after pediatric Emergencies (CAARE) — CAARE is a technology-enhanced stepped model of care that is designed to deliver education at the bedside to caregivers of children under age 12 years hospitalized for pediatric injury about mental health recovery after pediatric injury as well as risk assessment and brief intervention for high-risk patients (Step 1), foster symptom self-monitoring and reinforcement of coping skills via mHealth tools (Step 2), screen for caregivers' and children's PTSD and depression 30 days post-injury (Step 3), and provide a referral and warm hand-off to mental health services if needed (Step 4).
  Arms: Caregivers' Aid to Accelerate Recovery after pediatric Emergencies (CAARE)

SUMMARY:
Pediatric traumatic injury (PTI) is a public health priority, with more than 125,000 children experiencing injuries that require hospitalization each year. These children, and their caregivers, are affected in many ways that may affect quality of life, emotional and behavioral health, physical recovery, family roles and routines, and academic functioning; yet US trauma centers do not adequately address these outcomes and a scalable national model of care for these families is needed. This proposal builds on prior research from the investigative team to test a technology-assisted, stepped care behavioral health intervention for children (<12 years) and their caregivers after PTI, CAARE (Caregivers' Aid to Accelerate Recovery after pediatric Emergencies), via a hybrid type I effectiveness-implementation trial with 348 families randomly assigned to CAARE (n=174) vs. guideline-adherent enhanced usual care (EUC) (n=174).

DETAILED DESCRIPTION:
Annually, ~8 million children receive emergency care due to injury, over 125,000 of whom experience pediatric traumatic injury (PTI) - injuries so severe that they are hospitalized, typically after motor vehicle crashes, falls, animal attacks, gunshot wounds, or being struck by a car or other object. Roughly 1 in 3 develop posttraumatic stress disorder (PTSD) and/or depression after PTI - risk factors for poor physical recovery, social and school-related impairment, and disruption of roles and routines. Moreover, >50% of caregivers of children with PTI are highly distressed in the acute stages of recovery and themselves have high risk of PTSD and depression. This is concerning because caregivers' mental health is highly correlated with children's outcomes. Interventions that improve families' quality of life and emotional and behavioral recovery after PTI are a public health priority. However, trauma centers do not currently have best-practice interventions in place to address this need. Studies led by our team found that few Level 1 pediatric trauma centers have embedded behavioral health programs and that there is high interest in learning how to implement such programs. Many centers are eager to implement cost-efficient models of care. The 2022 American College of Surgeons guidelines explicitly recommend mental health intervention. Pediatric trauma centers therefore are ideally positioned and motivated to embed best-practice care to address the emotional and behavioral needs of children and families.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers (≥18 years old) of children hospitalized with pediatric injury
* Children hospitalized with pediatric injury <12 years old
* Screen positive on the ASC-Kids (aged 8-11 years) or PDI Caregiver measure of acute distress.

Exclusion Criteria:

* A caregiver whose primary language is not English
* A cognitive challenge (caregiver or child) that would impair ability to consent
* Presence of a self-afflicted injury
* Presence of injuries resulting from caregiver abuse or neglect (these patients will follow an alternative treatment path).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in scores in child self-report and caregiver proxy-report of child Quality of Life (QOL) | From enrollment (baseline) to 3-month, to 6-month, until end of treatment at 12-month
  PROMIS General Life Satisfaction (Caregiver QOL) consists of 10 items that assess general domains of health and functioning including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life. The Pediatric Quality of Life Inventory (PEDSQL) consists of 23 items in that comprise four Generic Core Scales: Physical Functioning (8 items), Emotional Functioning (5 items), Social Functioning (5 items), and School Functioning (5 items). Items on the PedsQL are reverse scored and transformed to a 0-100 scale. Higher scores indicate better health related quality of life.
Change in scores in caregiver self-report of PTSD | From 3-month, to 6-month, until end of treatment at 12-month
  The Abbreviated PTSD Checklist for DSM-5 (PCL-5) will be used to assess caregiver PTSD. The 20 items are rated on a scale from 0-4, with a total symptom severity score calculated by summing all item scores, resulting in a possible range of 0-80, with higher scores indicating the increase in severity of PTSD in caregivers.
Change in scores in caregiver self-report of caregiver depression | From 3-month, to 6-month, until end of treatment at 12-month
  Patient Health Questionnaire (PHQ-8) will be used to assess symptoms of caregiver depression, with scores ranging from 0-24 and higher scores indicating higher depression symptoms.
Change of child externalizing problems from 3 month to 12 month | From 3-month, to 6-month, until end of treatment at 12-month
  The investigators will use the BASC-3 Behavioral and Emotional Screening System (BESS) to assess children's externalizing behaviors using the BESS Externalizing Problems Composite scale via self-report (ages 6-11) and caregiver proxy report (ages 2-11). The BASC-3 Behavioral and Emotional Screening System (BESS) uses a Behavioral and Emotional Risk Index (BERI) T score to indicate a student's risk level for behavioral and emotional problems. Normal risk: 60 or lower, elevated risk: 61-70, extremely elevated risk: 71 or higher
Change in scores in child self-report and caregiver proxy-report of child PTSD | From 3-month, to 6-month, until end of treatment at 12-month
  The Child and Adolescent Trauma Screen (CATS) will be used to assess child PTSD via both self report (ages 7-11) and caregiver proxy report (ages 3-11). The CATS has 15 items measuring traumatic events, 20 items measuring DSM-5 PTSD symptoms, and 5 items measuring psychosocial functioning. Ages 3-6: The total symptom score is calculated by summing up the items 1-16 (possible range = 0-48), ≥ 16 is an indication of a clinically relevant level of symptoms. Ages 7-17: The total symptom score is calculated by summing up the raw scores of items 1-20 (possible range = 0-60), ≥ 21 as indication of a clinically relevant level of symptoms
Change in scores in child self-report (ages 6-11) of child depression | From 3-month, to 6-month, until end of treatment at 12-month
  The Center for Epidemiological Studies Depression Scale for Children (CESD) is a 20-item measure assessing depression in children ages 6-17. Scores range from 0-60, with higher scores indicating higher symptoms of depression in children

SECONDARY OUTCOMES:
Number of caregivers with service engagement | From 3-month, to 6-month, until end of treatment at 12-month
  Mental health care service engagement will be assessed using the National Health Injury Survey (NHIS) mental health service utilization items and also items assessing barriers to healthcare.
Mean number of child missed daycare/school days due to pediatric traumatic injury | At 3-month, 6-month, and 12-month
  Caregiver will report on children's number of school and/or daycare days missed due to the injury
Change in caregiver health status | From enrollment (baseline) to 3-month, to 6-month, to end of treatment at 12-month
  36-item Short Form Health Survey (SF-36) will be used to assess a generic indicator of caregivers' health status assessing physical health, role, social, and mental health function. Higher scores indicate more favorable health state, with scores ranging from 0-100.
Change in caregiver work and productivity status | From enrollment (baseline) to 3-month, to 6-month, to end of treatment at 12-month
  A single questionnaire item asking caregivers whether they are working, laid off/looking for work, not working and not searching for employment, a student, a homemaker, volunteering, caretaking for another, retired, hospitalized or in a skilled nursing facility, in jail, disabled, or homeless.
Number of children with service engagement | From 3-month, to 6-month, until end of treatment at 12-month
  Mental health care service engagement will be assessed using the National Health Injury Survey (NHIS) mental health service utilization items and also items assessing barriers to healthcare.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Ridings, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (4):
- United States (4):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kentucky Children's Hospital, Lexington, Kentucky
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Memorial Hermann Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided